CLINICAL TRIAL: NCT02391519
Title: Effects of High Altitude on 5' Adenosine Monophosphate-activated Protein Kinase (AMPK) Activation and Peroxisome Proliferator-activated Receptor Gamma (PPARγ) Regulation
Brief Title: Effects of High Altitude on AMPK Activation
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-2178
Record Dates: First submitted 2015-03-03; First posted 2015-03-18 (Estimated); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Pregnancy; IUGR; Preeclampsia
Keywords: Pregnancy; High altitude; vasoreactivity; myometrial arteries
MeSH Terms: conditions — Pre-Eclampsia; Altitude Sickness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Myometrial tissue, Cord Blood, Placental Tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High Altitude (3000 m): Collection of myometrial, cord blood, and placental tissue samples from women at high altitude (Summit County) and low altitude (Denver) in Colorado in order to determine if residence at altitude during pregnancy changes the vasoreactivity of myometrial arteries (MA).
  Interventions: Procedure: Collection of myometrial, cord blood, and placental tissue samples
- Low Altitude (1600 m): Collection of myometrial, cord blood, and placental tissue samples from women at high altitude (Summit County) and low altitude (Denver) in Colorado in order to determine if residence at altitude during pregnancy changes the vasoreactivity of myometrial arteries (MA).
  Interventions: Procedure: Collection of myometrial, cord blood, and placental tissue samples

INTERVENTIONS:
Procedure: Collection of myometrial, cord blood, and placental tissue samples — We propose to collect myometrial, cord blood, and placental tissue samples from women at high altitude (Summit County) and low altitude (Denver) in Colorado in order to determine if residence at altitude during pregnancy changes the vasoreactivity of myometrial arteries (MA).

SUMMARY:
Pregnancy elicits adaptive changes in uteroplacental blood flow, which are altered at high altitude and may contribute to the observed 3-fold increase in intrauterine growth restriction (IUGR) and preeclampsia (PreE). The investigators propose to collect myometrial, cord blood, and placental tissue samples from women at high altitude (Summit County) and low altitude (Denver) in Colorado in order to determine if residence at altitude during pregnancy changes the vasoreactivity of myometrial arteries (MA). If altered MA vasoreactivity is found, further studies may be able to link these changes to the increased rates of PreE and IUGR at altitude and contribute to the understanding of these two disorders.

DETAILED DESCRIPTION:
The Investigators will determine if residence at altitude during pregnancy changes the vasoreactivity of myometrial arteries. This will be novel information regarding pregnancy at altitude and of significance not just for women and families in Colorado, but also at high-altitude locations throughout the world. If altered MA vasoreactivity is found, further studies may be able to link these changes to the increased rates of PreE and IUGR at altitude and contribute to the understanding of these two disorders.

The Investigators will also determine whether the chronic hypoxia of high altitude alters DNA methylation patterns and expression of key genes involved in metabolic homeostasis in maternal, placental and fetal cells and, in turn, the relationship of these changes to fetal growth and maternal well-being.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for cesarean delivery at University of Colorado Hospital (Denver, 1600 m) and St. Anthony's Summit Medical Center (Summit County, 3000 m)
* Cesarean delivery at a prescheduled time without any labor, typically at 39 weeks gestation

Exclusion Criteria:

* Women will be excluded if there are co-existing medical diagnoses that are known to affect vascular parameters (i.e., diabetes mellitus, gestational diabetes, any hypertensive disorder of pregnancy, or a current smoker).
* Women with multiple gestations and preterm deliveries will also be excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women scheduled for cesarean delivery at University of Colorado Hospital (Denver, 1600 m) and St. Anthony's Summit Medical Center (Summit County, 3000 m) will be identified. In order to avoid any possible confounding effects of labor or prematurity, only women with elective cesarean deliveries will be approached for enrollment (cesarean delivery at a prescheduled time without any labor, typically at 39 weeks gestation).
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2016-01; Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Myometrial artery dimensions | Up to 1 year
  Myometrial artery dimensions as quantified by immunohistochemistry or other staining techniques, and results of studies of isolated myometrial artery studies in which vasoconstrictor and vasodilator responses to pharmacological agonists are measured using absolute values and the percent maximal contraction to potassium chloride.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Moore, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Background] Osol G, Moore LG. Maternal uterine vascular remodeling during pregnancy. Microcirculation. 2014 Jan;21(1):38-47. doi: 10.1111/micc.12080. PMID 23941526
- [Background] Zamudio S, Palmer SK, Droma T, Stamm E, Coffin C, Moore LG. Effect of altitude on uterine artery blood flow during normal pregnancy. J Appl Physiol (1985). 1995 Jul;79(1):7-14. doi: 10.1152/jappl.1995.79.1.7. PMID 7559250
- [Background] Krampl ER, Espinoza-Dorado J, Lees CC, Moscoso G, Bland JM, Campbell S. Maternal uterine artery Doppler studies at high altitude and sea level. Ultrasound Obstet Gynecol. 2001 Dec;18(6):578-82. doi: 10.1046/j.0960-7692.2001.00579.x. PMID 11844192
- [Background] Julian CG, Galan HL, Wilson MJ, Desilva W, Cioffi-Ragan D, Schwartz J, Moore LG. Lower uterine artery blood flow and higher endothelin relative to nitric oxide metabolite levels are associated with reductions in birth weight at high altitude. Am J Physiol Regul Integr Comp Physiol. 2008 Sep;295(3):R906-15. doi: 10.1152/ajpregu.00164.2008. Epub 2008 Jun 25. PMID 18579652
- [Background] Palmer SK, Moore LG, Young D, Cregger B, Berman JC, Zamudio S. Altered blood pressure course during normal pregnancy and increased preeclampsia at high altitude (3100 meters) in Colorado. Am J Obstet Gynecol. 1999 May;180(5):1161-8. doi: 10.1016/s0002-9378(99)70611-3. PMID 10329872
- [Background] Moore LG, Hershey DW, Jahnigen D, Bowes W Jr. The incidence of pregnancy-induced hypertension is increased among Colorado residents at high altitude. Am J Obstet Gynecol. 1982 Oct 15;144(4):423-9. doi: 10.1016/0002-9378(82)90248-4. PMID 7124861
- [Background] Jensen GM, Moore LG. The effect of high altitude and other risk factors on birthweight: independent or interactive effects? Am J Public Health. 1997 Jun;87(6):1003-7. doi: 10.2105/ajph.87.6.1003. PMID 9224184
- [Background] Keyes LE, Armaza JF, Niermeyer S, Vargas E, Young DA, Moore LG. Intrauterine growth restriction, preeclampsia, and intrauterine mortality at high altitude in Bolivia. Pediatr Res. 2003 Jul;54(1):20-5. doi: 10.1203/01.PDR.0000069846.64389.DC. Epub 2003 Apr 16. PMID 12700368
- [Background] White MM, McCullough RE, Dyckes R, Robertson AD, Moore LG. Chronic hypoxia, pregnancy, and endothelium-mediated relaxation in guinea pig uterine and thoracic arteries. Am J Physiol Heart Circ Physiol. 2000 Jun;278(6):H2069-75. doi: 10.1152/ajpheart.2000.278.6.H2069. PMID 10843906
- [Background] Xiao D, Longo LD, Zhang L. Role of KATP and L-type Ca2+ channel activities in regulation of ovine uterine vascular contractility: effect of pregnancy and chronic hypoxia. Am J Obstet Gynecol. 2010 Dec;203(6):596.e6-12. doi: 10.1016/j.ajog.2010.07.038. PMID 20817142
- [Background] Luksha L, Luksha N, Kublickas M, Nisell H, Kublickiene K. Diverse mechanisms of endothelium-derived hyperpolarizing factor-mediated dilatation in small myometrial arteries in normal human pregnancy and preeclampsia. Biol Reprod. 2010 Nov;83(5):728-35. doi: 10.1095/biolreprod.110.084426. Epub 2010 Jul 7. PMID 20610807
- [Background] Cockell AP, Poston L. Flow-mediated vasodilatation is enhanced in normal pregnancy but reduced in preeclampsia. Hypertension. 1997 Aug;30(2 Pt 1):247-51. doi: 10.1161/01.hyp.30.2.247. PMID 9260988
- [Background] Sladek SM, Magness RR, Conrad KP. Nitric oxide and pregnancy. Am J Physiol. 1997 Feb;272(2 Pt 2):R441-63. doi: 10.1152/ajpregu.1997.272.2.R441. PMID 9124465
- [Background] Clapp JF 3rd, Capeless E. Cardiovascular function before, during, and after the first and subsequent pregnancies. Am J Cardiol. 1997 Dec 1;80(11):1469-73. doi: 10.1016/s0002-9149(97)00738-8. PMID 9399724
- [Background] Palmer SK, Zamudio S, Coffin C, Parker S, Stamm E, Moore LG. Quantitative estimation of human uterine artery blood flow and pelvic blood flow redistribution in pregnancy. Obstet Gynecol. 1992 Dec;80(6):1000-6. PMID 1448242
- [Background] Kametas NA, McAuliffe F, Krampl E, Chambers J, Nicolaides KH. Maternal cardiac function during pregnancy at high altitude. BJOG. 2004 Oct;111(10):1051-8. doi: 10.1111/j.1471-0528.2004.00246.x. PMID 15383106
- [Background] Zamudio S, Palmer SK, Dahms TE, Berman JC, Young DA, Moore LG. Alterations in uteroplacental blood flow precede hypertension in preeclampsia at high altitude. J Appl Physiol (1985). 1995 Jul;79(1):15-22. doi: 10.1152/jappl.1995.79.1.15. PMID 7559213
- [Background] Mateev S, Sillau AH, Mouser R, McCullough RE, White MM, Young DA, Moore LG. Chronic hypoxia opposes pregnancy-induced increase in uterine artery vasodilator response to flow. Am J Physiol Heart Circ Physiol. 2003 Mar;284(3):H820-9. doi: 10.1152/ajpheart.00701.2002. Epub 2002 Nov 14. PMID 12433660
- [Background] Wang X, Proud CG. The mTOR pathway in the control of protein synthesis. Physiology (Bethesda). 2006 Oct;21:362-9. doi: 10.1152/physiol.00024.2006. PMID 16990457